CLINICAL TRIAL: NCT00248131
Title: An Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of Octreotide Acetate in Microspheres in the Therapy of Patients With Moderately Severe or Severe Non-proliferative Diabetic Retinopathy (NPDR) or Low Risk Proliferative Diabetic Retinopathy (PDR)
Brief Title: Extension Study of Long-term Safety and Tolerability of Octreotide Acetate in Patients With Moderately Severe or Severe Non-proliferative Diabetic Retinopathy or Low Risk Proliferative Diabetic Retinopathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMS9950802E1
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic retinopathy, octreotide acetate in microspheres
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Octreotide; Microspheres

INTERVENTIONS:
Drug: Octreotide acetate in microspheres

SUMMARY:
This multicenter, open-label extension study will evaluate the long-term tolerability and safety for patients completing study CSMS995 0802. During this extension study, all patients will receive open-label treatment of octreotide acetate in microspheres every 4 weeks for 2 years for the treatment of moderately severe to severe NPDR and low risk PDR.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent provided prior to participation in the extension study
* successful completion of study CSMS995 0802
* willingness to comply with all study requirements

Exclusion Criteria:

* more than 8 weeks interval since the completion of study CSMS995 0802
* premature discontinuation from study CSMS995 0802

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2005-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
long-term safety and tolerability

SECONDARY OUTCOMES:
monitor long-term efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals